CLINICAL TRIAL: NCT01174355
Title: A Multicenter, Open Label, Escalating Dose Study to Assess the Tolerability and the Safety and to Explore the Efficacy and the Pharmacokinetics of ND0801 in Adult Patients With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Study of ND0801 in Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ND0801/001
Record Dates: First submitted 2010-08-01; First posted 2010-08-03 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Attention Deficit and Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ND0801 (Experimental)
  Interventions: Drug: ND0801

INTERVENTIONS:
Drug: ND0801 — Confidential

SUMMARY:
A multicenter, open label, escalating dose study to assess the tolerability and the safety and to explore the efficacy and the pharmacokinetics of ND0801 in adult patients with attention deficit/hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Men and women 18-55 years of age.
* Primary DSM-IV diagnosis of adult ADHD confirmed by senior physician
* Capable and willing to provide informed consent
* Able to adhere to the treatment schedule, and withdrawal of ongoing pharmacotherapy for the treatment of ADHD prior to the beginning of the study treatment and during the study drug treatment.
* Subjects must be able to read, hear, write and speak the local language.
* Subject has signed a written informed consent to participate in the study.

Exclusion Criteria:

* Unstable or significant medical disorder.
* Current (within 12 months of baseline) primary or secondary depression.
* History of substance abuse or dependence within the past 6 months
* Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features
* Bipolar disorder
* Eating disorder
* Obsessive compulsive disorder
* Post-traumatic stress disorder
* Current generalized anxiety disorder
* Presence of a personality disorder
* Individuals with a significant other neurological disorder.
* Use of any investigational drug within 4 weeks of the randomization visit
* Known or suspected pregnancy
* Women who are breast-feeding
* Women of childbearing potential and not using a medically accepted form of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability Evaluation | 1 week
  Safety and tolerability of ND0801 will be based on adverse events reporting by the subjects during the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rambam Hospital, Haifa
  - Shalvata Mental Health Center (SMHC), Hod HaSharon